CLINICAL TRIAL: NCT04336995
Title: Echocardiographic Assessment of Pulmonary Transit Time Following Exercise
Brief Title: Exercise Pulmonary Transit Time
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Ken Monahan, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB200429
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Results first posted 2022-07-12 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure, Diastolic
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — Echocardiography

STUDY DESIGN:
Intervention Model Description: small pilot study to test technical feasibility
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Exercise (Other): Everyone is in this arm
  Interventions: Diagnostic Test: contrast echocardiography

INTERVENTIONS:
Diagnostic Test: contrast echocardiography — giving echocardiographic contrast and taking echocardiographic images before and after exercise

SUMMARY:
The study seeks to measure pulmonary transit time via contrast-echocardiography before and after exercise.

DETAILED DESCRIPTION:
The ability to measure the amount of blood in the lungs using heart-ultrasound (echocardiography) can be useful to estimate how much fluid is in a patient's circulation, which can influence diagnosis and treatment of certain types of heart failure. In some patients, the amount of fluid is normal at rest, but can increase with activity and thus a diagnosis of heart failure can only be made after exercising. Currently, the amount of fluid is measured invasively. We have shown that echocardiography can measure the amount of fluid in the lung circulation at rest without the need for an invasive procedure. We now seek to find out if we can make a similar measurement after exercise. If successful, the need for catheter procedures may be reduced in certain types of heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Able to give informed consent

Exclusion Criteria:

1. Known allergic reaction to Definity or Optison ultrasound contrast
2. Pregnancy/Nursing - as assessed/disclosed by the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ken Monahan, MD, Principal Investigator — VUMC
Locations (1):
- VHVI, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercise
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Exercise
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Pulmonary Transit Time
Description: interval required for the pulmonary blood volume to traverse the pulmonary circulation
Time Frame: 3-10 seconds
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Exercise
Number analyzed (Participants) | 14
seconds | 2.5 (0.5)

ADVERSE EVENTS:
Time Frame: day of study
Arm/Group | Exercise
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT04336995/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/95/NCT04336995/ICF_001.pdf